CLINICAL TRIAL: NCT01791361
Title: Medical Records Review to Describe the Patterns of KRAS Testing and Vectibix Use in Europe
Status: Completed | Type: Observational
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Other Study IDs: 20101120
Record Dates: First submitted 2012-06-05; First posted 2013-02-15 (Estimated); Last update posted 2022-09-10 (Actual); Status verified 2022-09

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Round 1: 50 oncologists participate in Round 1. At least 3 medical records will be reviewed per oncologist
  Interventions: Other: Other
- Round 2: 50 oncologists will participate in Round 2. At least 3 medical records will be reviewed per oncologist. Round 2 will occur approximately 12 months after Round 1
  Interventions: Other: Other
- Round 3: 50 oncologists will participate in Round 3. At least 3 medical records will be reviewed per oncologist. Round 3 will occur approximately 24 months after Round 1
  Interventions: Other: Other

INTERVENTIONS:
Other: Other — No intervention other than routine medical care
  Other Names: Medical Records Review

SUMMARY:
This non-interventional retrospective medical record review study will assess the prevalence of KRAS testing and the impact of the KRAS test result on patterns of Vectibix use in patients with metastatic colorectal cancer (mCRC) treated with Vectibix in selected European countries over 3 rounds. As the optimal use of Vectibix also requires accurate KRAS mutation testing, this study will also assess data from the laboratory that performed the KRAS test. The study will also monitor changes in the pattern of Vectibix treatment between the different rounds of the study.

DETAILED DESCRIPTION:
The medical record review will be conducted for 3 rounds in months 0, 12, and 24 after the first medical record abstraction. Before the beginning of the study, a sampling list will be created by Amgen by merging lists of oncologists (and their contact information) to be collected from Cegedim, the ESMO, from major cancer centers and oncology clinics in various countries within Europe. In each round of medical record review, potential participating oncologists will be randomly sampled from all identified oncologists. Potential oncologists will be contacted by letter, telephone or email. The oncologists will be introduced to the study, and their eligibility to participate in the study will be assessed using a standardized questionnaire. The number of oncologists sampled per country will be proportional to the number of oncology centers per country. Approximately 50 oncologists will participate in each round of the study. From each eligible participating oncologist, study staff will then obtain approximately 3 or more medical records for patients who have received Vectibix for the treatment of mCRC during the 6-month period prior to the time of contact with the relevant oncologist and are not involved in an experimental clinical trial when treated with Vectibix. A written consent may be obtained from participating patients to access their medical records, depending on local laws. Medical information will be abstracted from the medical records using standardized forms. Such medical information will include the occurrence and timing of treatment with Vectibix and oxaliplatin-containing chemotherapy, diagnosis of mCRC and the occurrence, timing and results of KRAS testing. The oncologist will also be asked to collect information from the pathology laboratory that performed the KRAS mutation test on the patient, using a standardized pathology data extraction form.

ELIGIBILITY:
Physician Inclusion Criteria:

* Must be a practicing oncology specialist
* Must treat at least 5 new or continuing patients with metastatic colorectal cancer per quarter
* Must have prescribed Vectibix to treat at least 5 new or continuing patients with metastatic colorectal cancer in the past 6 months

Physician Exclusion Criteria:

* Must be the only oncologist sampled at the same medical centre for that round of the study
* Must not have taken part in the study previously

Patient Inclusion Criteria

* Must have received Vectibix for the treatment of metastatic colorectal cancer during the 6-month period prior to the time when medical records are obtained
* Must not have been in any experimental clinical trial at the time of receiving Vectibix
* Must provide written consent to allow access to their medical records (if local laws require it)
* Must not have taken part in the study before

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oncologists satisfying all of the physician eligibility criteria will be eligible to participate in the medical records review study. From each eligible oncologist, medical records from 3 or more patients who satisfy all the patient inclusion criteria will be obtained.
Sampling Method: Probability Sample
Enrollment: 439 (Actual)
Dates: Start 2012-09-19 (Actual); Primary Completion 2015-06-02 (Actual); Study Completion 2015-06-02 (Actual)

PRIMARY OUTCOMES:
The prevalence of KRAS testing and impact of the KRAS test results on patterns of Vectibix use in patients with metastatic colorectal cancer (mCRC) treated with Vectibix | 3 years
  The proportion of patients with mCRC treated with Vectibix only or treated with Vectibix and concurrently treated with oxaliplatin-containing chemotherapy who received a KRAS test to determine tumor KRAS status prior to treatment with Vectibix, and characterize the results of above testing for KRAS testing: proportion that are mutant, wild-type or unknown but tested

SECONDARY OUTCOMES:
The proportion of oncologists who agree to participate in the study | 3 years
The proportion of oncologists that conduct a KRAS testing prior to Vectibix prescription in patients with mCRC treated with Vectibix | 3 years
The proportion of laboratories that participate in the European Society of Pathology (ESP) Quality Assurance Scheme or are certified by an ESP approved accreditation body | 3 years
  The study will obtain data from laboratories that tested KRAS status on mCRC patients who were treated with Vectibix.
The proportion of laboratories that use a CE-marked or otherwise validated KRAS detection method | 3 years
  The study will obtain data from laboratories that tested KRAS status on mCRC patients who were treated with Vectibix.
To characterize the results of KRAS testing in the three rounds of chart abstraction that will be carried out at 0, 12 and 24 months to indicate if there are any differences in results from each of the three rounds | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (80):
- Belgium (6):
  - Research Site, Bonheiden
  - Research Site, Brasschaat
  - Research Site, Bruges
  - Research Site, Haine Saint Paul - La Louviere
  - Research Site, Liège
  - Research Site, Merksem
- Czechia (6):
  - Research Site, Brno
  - Research Site, Chomutov
  - Research Site, Jihlava
  - Research Site, Pilsen
  - Research Site, Prague
  - Research Site, Ústí nad Labem
- Denmark (4):
  - Research Site, Copenhagen
  - Research Site, Esbjerg
  - Research Site, Herning
  - Research Site, Hillerød
- France (19):
  - Research Site, Ajaccio
  - Research Site, Avignon
  - Research Site, Bordeaux
  - Research Site, Brest
  - Research Site, Clermont-Ferrand
  - Research Site, Évry
  - Research Site, Grenoble
  - Research Site, La Tronche
  - Research Site, Limoges
  - Research Site, Lyon
  - Research Site, Marseille
  - Research Site, Muret
  - Research Site, Nancy
  - Research Site, Perpignan
  - Research Site, Périgueux
  - Research Site, Reims
  - Research Site, Saint-Grégoire
  - Research Site, Strasbourg
  - Research Site, Toulouse
- Germany (21):
  - Research Site, Ahaus
  - Research Site, Amberg
  - Research Site, Arnsberg
  - Research Site, Aschersleben
  - Research Site, Bonn
  - Research Site, Cologne
  - Research Site, Dessau
  - Research Site, Duisburg
  - Research Site, Frankfurt am Main
  - Research Site, Goslar
  - Research Site, Halle
  - Research Site, Hamburg
  - Research Site, Leipzig
  - Research Site, Leverkusen
  - Research Site, München
  - Research Site, Osnabrück
  - Research Site, Pforzheim
  - Research Site, Recklinghausen
  - Research Site, Regensburg
  - Research Site, Saarbrücken
  - Research Site, Wilhelmshaven
- Italy (7):
  - Research Site, Foggia
  - Research Site, Legnago VR
  - Research Site, Napoli
  - Research Site, Ravenna
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Vimercate MB
- Netherlands (3):
  - Research Site, Amstelveen
  - Research Site, Doetinchem
  - Research Site, Eindhoven
- Spain (9):
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, Bilbao, Basque Country
  - Research Site, Burgos, Castille and León
  - Research Site, Granollers, Catalonia
  - Research Site, Ourense, Galicia
  - Research Site, Pamplona, Navarre
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Castellon, Valencia
  - Research Site, Madrid
- Sweden (5):
  - Research Site, Eskilstuna
  - Research Site, Gothenburg
  - Research Site, Karlskrona
  - Research Site, Skövde
  - Research Site, Västerås

REFERENCES:
- [Background] Han van Krieken J, Kafatos G, Bennett J, Mineur L, Tomasek J, Rouleau E, Fabian P, De Maglio G, Garcia-Alfonso P, Aprile G, Parkar P, Downey G, Demonty G, Trojan J. Panitumumab use in metastatic colorectal cancer and patterns of RAS testing: results from a Europe-wide physician survey and medical records review. BMC Cancer. 2017 Nov 28;17(1):798. doi: 10.1186/s12885-017-3740-4. PMID 29183279
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com